CLINICAL TRIAL: NCT01133925
Title: Optical Coherence Tomography in Long Native Coronary Artery Lesions Treated With Multiple Novel Zotarolimus-eluting Stents: LONG OCT STUDY
Brief Title: Optical Coherence Tomography in Long Lesions
Acronym: LONG OCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Case Western Reserve University (Other); Medtronic Vascular (Industry)
Responsible Party: Giulio Guagliumi, Cardiovascular Department Ospedali Riuniti di Bergamo, Italy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-003-08
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Drug Eluting Stent; Optical Coherence Tomography; Thrombosi; Long lesions in native vessels requiring overlap
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ODESSA (Active Comparator): ODESSA trial (NCT 00693030)Patients were randomized (2:2:2:1) to receive multiple TAXUS Libertè™ vs Cypher Select™ vs Endeavor™ vs Libertè BM stents, in overlap. At 6-months follow-up coronary angiography (QCA), IVUS and Optical Coherence Tomography assessments were made. Data reported in J. Am. Coll. Cardiol. Intv. 2010;3;531-539. DOI 10.1016/j.jcin.2010.02.008.
  Interventions: Device: Sirolimus Eluting Stent; Device: Paclitaxel Eluting Stent; Device: Zotarolimus eluting stent
- Resolute Sprint arm (Experimental): Zotarolimus Eluting stents (Resolute Sprint) implanted in overlap to treat long coronary lesions
  Interventions: Device: Resolute Sprint

INTERVENTIONS:
Device: Resolute Sprint — Zotarolimus Eluting Stent (Resolute Sprint) implanted in overlap
  Arms: Resolute Sprint arm
Device: Sirolimus Eluting Stent — Cypher stents implanted in overlap
  Arms: ODESSA
Device: Paclitaxel Eluting Stent — Taxus stents implanted in overlap
  Arms: ODESSA
Device: Zotarolimus eluting stent — Endeavor stents implanted in overlap
  Arms: ODESSA

SUMMARY:
Increasing lesion complexity in percutaneous coronary interventions (PCI) has warranted the use of overlapping drug-eluting stents. Whether the substantial impairment of arterial healing observed at sites of overlap in preclinical pathologic studies persists in patients undergoing PCI is unknown. Consecutive patients with long lesions in native coronary vessels requiring stents in overlap are prospectively assigned to receive multiple zotarolimus eluting stents (Resolute Sprint). The completeness of stent struts coverage and/or late malapposition are evaluated by Optical Coherence Tomography at 6 months follow-up.Data will be compared to the historical arm of ODESSA trial (patients treated with multiple sirolimus-,paclitaxel polymer-or zotarolimus eluting stents).

DETAILED DESCRIPTION:
It is not unknown whether overlapping drug-eluting stents provide increased vessel toxicity. Given the association of delayed healing and incomplete endothelialization observed in animal and human autopsy studies at overlapping sites it is unclear why most patients do well with multiple DES implanted. OCT detects smaller degrees of in-stent neointima more accurately than IVUS and might be a useful method for identify strut coverage and/or malapposition.

Patients if eligible on the basis of clinical and angiographic criteria, are assigned to receive multiple Resolute Sprint™. Stent implantation are done accordingly to the normal interventional practice. QCA and IVUS are performed at the end of optimal stents placement per visual judgement (residual stenosis < 10%, TIMI 3 flow). Stent, lumen size and volume as well as complete stent strut apposal will be determined by IVUS analysis. Clinical follow-up will take place at 1 month (±1 week), 6 months (±2 weeks) and 1 year (±2 weeks). At 6-months follow-up all patients will undergo a quantitative coronary angiography (QCA), IVUS and Optical Coherence Tomography (LightLab OCT Imaging M2, automated pull back and flushing combination)assessments.

OCT images will be acquired at 15-30 frames per second. Blind corelab quantitative strut by strut analysis will be performed using a novel dedicated software at each 0.5 mm section. The following OCT variables will be evaluated:number of visualized strut per section, mean-max neointimal thickness per section, % struts well apposed with neointima at overlapping vs non overlapping sites, % struts without neointima, % struts malapposed, rate of > 30% uncovered struts/total number of struts per section.

Obtained data will be compared with the data from a historical comparator (ODESSA trial that presented results from TAXUS Libertè™ vs Cypher Select™ vs Endeavor™ stents implanted in overlap to treat long lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia)
* Native coronary artery disease with >75% diameter stenosis (no prior stent implant, no prior brachytherapy)
* Lesion length > 20 mm
* Vessel size between 2.5 and 3.5 mm
* Multiple, overlapped Endeavor Resolute stents placement (intention to overlap > 4 mm).

Exclusion Criteria:

* Left main coronary artery disease
* Lesions in coronary artery bypass grafts
* Acute myocardial infarction
* Killip class IV
* Recent major bleeding (6 months)
* Renal failure with creatinine value > 2.5 mg/dl
* Left ventricular global ejection fraction ≤ 30%.
* Allergy to aspirin and or clopidogrel/ticlopidine
* Patient in anticoagulant therapy
* No suitable anatomy for OCT scan: (only ostial location, very tortuous anatomy, very distal or large vessels [> 3.5 mm in diameter])
* Target lesion(s) located in a major epicardial vessel or a side branch that has been previously treated with any type of percutaneous intervention (e.g., balloon angioplasty, cutting balloon, atherectomy) < 9 months prior to index procedure
* Target lesion restenotic from previous stent implantation
* Any lesion (target or non-target) that has been previously treated with brachytherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
In stent NIH at overlapping vs non overlapping sites | 6 month
  In-stent neointimal hyperplasia (NIH) thickness at 6 months, as measured by OCT, at overlapping vs non overlapping sites: superiority of Endeavor Resolute stent compared to Endeavor Sprint
Percent uncovered and malapposed struts in OCT | 6 month
  Proportion of stent struts uncovered and/or malapposed at 6 months, as measured by OCT, at overlapping vs non overlapping sites: non inferiority of Endeavor Resolute compared to Endeavor Sprint.

SECONDARY OUTCOMES:
Rate of > 30% uncovered struts/total number of struts per section. | 6 months
MACE Rates | 1-6 and 12 months
  All specific components of MACE (cardiac death, myocardial infarction (Q wave and non Q wave), and target vessel revascularization) will be summarized. MACE shall be assessed at, discharge (or within 7 days, whichever comes first), 1, 6 and 12 months post index procedure.
IVUS parameters | 6 months
  Based on IVUS Core Lab analysis including:
  * Neointimal volume, stent volume, lumen volume and percent net volume obstruction
  * Neointimal Thickness: Neointimal hyperplasia (NIH) inside all struts (mean, median, max)
  * Percent NIH Area= ([stent area-lumen area]/stent area) X 100
  * Rate of > 30% uncovered struts/total number of struts per section.
QCA Parameters | 6 months
  Based on Angiographic Core Lab analysis utilizing Quantitative Coronary Angiography (QCA) including:
  Mean lumen diameter, acute gain, late loss through 6 months, and binary restenosis (≥ 50% diameter stenosis) rate at 6 months post index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — Cardiovascular Department Ospedali Riuniti di Bergamo
Locations (1):
- Cardiovascular Department Ospedali Riuniti di Bergamo, Bergamo, BG, Italy

REFERENCES:
- [Background] Guagliumi G, Musumeci G, Sirbu V, Bezerra HG, Suzuki N, Fiocca L, Matiashvili A, Lortkipanidze N, Trivisonno A, Valsecchi O, Biondi-Zoccai G, Costa MA; ODESSA Trial Investigators. Optical coherence tomography assessment of in vivo vascular response after implantation of overlapping bare-metal and drug-eluting stents. JACC Cardiovasc Interv. 2010 May;3(5):531-9. doi: 10.1016/j.jcin.2010.02.008. PMID 20488410
- [Derived] Guagliumi G, Ikejima H, Sirbu V, Bezerra H, Musumeci G, Lortkipanidze N, Fiocca L, Tahara S, Vassileva A, Matiashvili A, Valsecchi O, Costa M. Impact of drug release kinetics on vascular response to different zotarolimus-eluting stents implanted in patients with long coronary stenoses: the LongOCT study (Optical Coherence Tomography in Long Lesions). JACC Cardiovasc Interv. 2011 Jul;4(7):778-85. doi: 10.1016/j.jcin.2011.04.007. PMID 21777886